CLINICAL TRIAL: NCT02846194
Title: Effects of Brief Guided Imagery for Chronic Pain in Patients Diagnosed With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pablo Roitman (Other)
Responsible Party: Sponsor-Investigator, Pablo Roitman, MD, Clalit Health Services
Organization: Clalit Health Services (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0015-16COM2
Record Dates: First submitted 2016-07-19; First posted 2016-07-27 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Fibromyalgia; Chronic Pain
Keywords: Fibromyalgia; Guided Imagery; chronic pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- brief guided imagery (Experimental): The study group of our research will go through six Brief Guided Imagery sessions. These sessions will be completed within two months and will last one hour each.
  Interventions: Behavioral: brief guided imagery
- control group (No Intervention)

INTERVENTIONS:
Behavioral: brief guided imagery
  Arms: brief guided imagery

SUMMARY:
The purpose of this study is to determine the effect that the Brief Guided Imagery (BGI) technique has on fibromyalgia patients suffering from chronic pain in regards to their sense of pain, wellbeing and quality of life.

This study will explore whether daily training of one to two minutes exercises in Brief Guided Imagery can reduce chronic pain and improve the quality of life of patients by studying specifically patients suffering from fibromyalgia.

Chronic pain is a common condition which affects person's physical and mental health. It occurs in between 10% to 40% of the population, depending on the exact research and chosen sample. In 2010 Manchikant et al. found an effect chronic pain has on human functioning and quality of life.

A research from 2007 defined chronic pain as pain that lasts more than three months. Being long lasting by its nature, chronic pain has an ongoing effect on deteriorating the quality of life. In this regards, quality of life is scientifically determined by five modes: i. Physical wellbeing. ii. Mental wellbeing. iii. Social wellbeing. iv. Emotional wellbeing, and v. sense of development and self-realization.

Chronic pain damages daily ongoing functions and is also related to sleep disturbances, stress and unemployment. A direct correlation was also found between chronic pain and psycho-social .

One of the many results of chronic pain is the huge impact on the economy, such as absence from work due to sick leaves. The overall cost of chronic pain was found to be one percent of the total expense on health. The frequency and impact of chronic pain is such that some professionals define it as an epidemic.

In many cases, chronic pain occurs with patients suffering from a wide spectrum of medical disorders. In 2007 Tunks et al. demonstrated that chronic pain often accompanies an illness that involves also a psychological aspect.

Both Baird et al. in 2004 and Menzies et al. in 2012 found a significant positive effect daily guided imagery exercises have on chronic pain. The study proposes to research the specific technique of Brief Guided Imagery on chronic pain, and will focus on patients suffering from fibromyalgia.

Fibromyalgia is a syndrome where a patient suffers from both chronic pain and a fatigue. The pain of fibromyalgia is characterized as abstract and non-localized, while the fatigue appears in a varying range of intensity. These symptoms are often accompanied by exhaustion, lack of energy, somatic disorders and psychologic symptoms such as depression.

The ongoing pain, fatigue and depression cause fibromyalgia patients to further suffer from sleep disorders and diminishing ability to function. Menzies et al. studied in 2012 the effect of guided imagery exercises on the stress level, pain, fatigue and depression. The study also examined different physiologic blood markers (such as proteins, cytokines and C reactive.

Menzies found a positive and significantly large improvement in the ability to control both stress and pain levels, and treat the depression of the participants. However, no significant changes were observed in the blood tests monitoring the levels of physiologic markers in the blood.

DETAILED DESCRIPTION:
Hypothesis Chronic pain imposes great suffering on patients as well as a heavy extra expenditure on the healthcare system . In addition, it many patients of chronic pain were found to also suffer from depression .

Guided imagery was found to be an effective technique to reduce chronic pain deriving from muscle or skeletal pain and from fibromyalgia. Guided imagery treatment carries low therapeutic costs and is noninvasive. It also puts the main emphasis of the process on the patient's satisfaction .Furthermore, a quantitative study by Kaplan et al. in 2014 found that daily exercises of guided imagery improved the sense of wellbeing among university students.

However, the improvement in the sense of wellbeing due to the practice of daily guided imagery was not tested empirically. Therefore, the investigators suggested research will look into the empirical effect of Brief Guided Imagery on chronic pain. The investigators will study the Colette technique for Brief Guided Imagery using short one to two minutes guided imagery exercises to try and determine the empiric effect brief exercises have on pain sensation and quality of life when performed by fibromyalgia patients with chronic pain.

ELIGIBILITY:
Inclusion Criteria:

* patient with Fibromyalgia that suffers from pain at least for 3 months

Exclusion Criteria:

* lliterates

Ages: 22 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-07; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Changes in Pain | Week 0 , Week 6
  pain will be measure by BPI questionnaire

SECONDARY OUTCOMES:
Changes in Quality of Life | week 0, Week 6
  Quality of Life will be measure by SF36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Anat Kaplun, Study Director — Ministry of Health, Israel; Pablo Roitman, MD, Principal Investigator — Clalit Heath Services
Locations (1):
- Ramat Eshkol Clalit health services, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Baird CL, Sands L. A pilot study of the effectiveness of guided imagery with progressive muscle relaxation to reduce chronic pain and mobility difficulties of osteoarthritis. Pain Manag Nurs. 2004 Sep;5(3):97-104. doi: 10.1016/j.pmn.2004.01.003. PMID 15359221
- [Background] Breivik H, Collett B, Ventafridda V, Cohen R, Gallacher D. Survey of chronic pain in Europe: prevalence, impact on daily life, and treatment. Eur J Pain. 2006 May;10(4):287-333. doi: 10.1016/j.ejpain.2005.06.009. Epub 2005 Aug 10. PMID 16095934
- [Background] Carlsson AM. Assessment of chronic pain. I. Aspects of the reliability and validity of the visual analogue scale. Pain. 1983 May;16(1):87-101. doi: 10.1016/0304-3959(83)90088-X. PMID 6602967
- [Background] Chandra A, Ozturk A. Quality of life issues and assessment tools as they relate to patients with chronic nonmalignant pain. Hosp Top. 2005 Winter;83(1):33-7. doi: 10.3200/htps.83.1.33-37. No abstract available. PMID 16092637
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Felce D, Perry J. Quality of life: its definition and measurement. Res Dev Disabil. 1995 Jan-Feb;16(1):51-74. doi: 10.1016/0891-4222(94)00028-8. PMID 7701092
- [Background] Richter K, Egger R, Negri L, Corsi R, Severini C, Kreil G. cDNAs encoding [D-Ala2]deltorphin precursors from skin of Phyllomedusa bicolor also contain genetic information for three dermorphin-related opioid peptides. Proc Natl Acad Sci U S A. 1990 Jun;87(12):4836-9. doi: 10.1073/pnas.87.12.4836. PMID 2352951
- [Background] Jain S, McMahon GF, Hasen P, Kozub MP, Porter V, King R, Guarneri EM. Healing Touch with Guided Imagery for PTSD in returning active duty military: a randomized controlled trial. Mil Med. 2012 Sep;177(9):1015-21. doi: 10.7205/milmed-d-11-00290. PMID 23025129
- [Background] Twycross A. Nurses' views about the barriers and facilitators to effective management of pediatric pain. Pain Manag Nurs. 2013 Dec;14(4):e164-e172. doi: 10.1016/j.pmn.2011.10.007. Epub 2011 Dec 14. PMID 24315269
- [Background] Lahmann C, Nickel M, Schuster T, Sauer N, Ronel J, Noll-Hussong M, Tritt K, Nowak D, Rohricht F, Loew T. Functional relaxation and guided imagery as complementary therapy in asthma: a randomized controlled clinical trial. Psychother Psychosom. 2009;78(4):233-9. doi: 10.1159/000214445. Epub 2009 Apr 28. PMID 19401624
- [Background] Lyon D, McCain N, Elswick RK, Sturgill J, Ameringer S, Jallo N, Menzies V, Robins J, Starkweather A, Walter J, Grap MJ. Biobehavioral examination of fatigue across populations: report from a P30 Center of Excellence. Nurs Outlook. 2014 Sep-Oct;62(5):322-31. doi: 10.1016/j.outlook.2014.06.008. Epub 2014 Jul 18. PMID 25218081
- [Background] D'Antoni ML, Harvey PL, Fried MP. Alternative medicine: does it play a role in the management of voice disorders? J Voice. 1995 Sep;9(3):308-11. doi: 10.1016/s0892-1997(05)80239-5. PMID 8541975
- [Background] McHorney CA, Haley SM, Ware JE Jr. Evaluation of the MOS SF-36 Physical Functioning Scale (PF-10): II. Comparison of relative precision using Likert and Rasch scoring methods. J Clin Epidemiol. 1997 Apr;50(4):451-61. doi: 10.1016/s0895-4356(96)00424-6. PMID 9179104
- See also: Prediction of function in daily life following multidisciplinary rehabilitation for individuals with chronic musculoskeletal pain; a prospective study — http://bmcmusculoskeletdisord.biomedcentral.com/articles/10.1186/1471-2474-8-65